CLINICAL TRIAL: NCT06626581
Title: A Cross-sectional Study on Iodine Status and Characteristics of Papillary Thyroid Cancer
Brief Title: Iodine Status and Characteristics of Papillary Thyroid Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Hai-qing Zhang, Chief physician, Shandong Provincial Hospital
Other Study IDs: ShandongPH 20240923
Record Dates: First submitted 2024-09-25; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: iodine status; papillary thyroid carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collect thyroid surgery specimens, serum, and urine from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Excessive iodine group: Residents with papillary thyroid cancer who have lived in excessive iodine areas for a long time (5 years or more). According to the report of Shandong linstitute of Endemic Disease Prevention and Control, three sub centers were selected in excessive iodine group(Jining/Liaocheng/Heze).
  Interventions: Dietary Supplement: Iodine excess
- Suitable iodine group: Residents with papillary thyroid cancer who have lived in suitable iodine areas for a long time (5 years or more). According to the report of Shandong linstitute of Endemic Disease Prevention and Control, three sub centers were selected in suitable iodine group(Jinan/Shenyang/Haerbin).
  Interventions: Dietary Supplement: Iodine suitable

INTERVENTIONS:
Dietary Supplement: Iodine excess — Iodine excess areas: water iodine ≥100μg/L; or urinary iodine concentration(median urinary iodine levels in children aged 8-10 years old) ≥300μg/L
  Groups: Excessive iodine group
Dietary Supplement: Iodine suitable — Iodine suitable areas: water iodine ≥40μg/L and ≤100μg/L; or urinary iodine concentration(median urinary iodine levels in children aged 8-10 years old) 100-199μg/L.
  Groups: Suitable iodine group

SUMMARY:
The effect of iodine on papillary thyroid cancer has been controversial for many years. The investigators designed a cross-sectional study and aimed to explore the relationship between the serum and urine iodine levels and the clinical and molecular characteristics of papillary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18~65 years old, gender not limited;
* Living in the residential area for at least 5 years;
* Patients diagnosed clinically with thyroid cancer and scheduled for thyroid surgery, with pathological diagnosis of papillary thyroid cancer;
* Complete clinical data: including general information, relevant laboratory tests, pathological reports, surgical reports, ultrasound reports, etc.

Exclusion Criteria:

* Pathological diagnosis of other types of thyroid cancer;
* Diagnosed with other types of cancer;
* There are serious comorbidities of the heart, liver, and kidneys;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three sub centers will be selected in high iodine areas (Jining, Liaocheng, Heze) and moderate iodine areas (Jinan, Shenyang, Harbin) respectively. People who have lived in these areas for more than 5 years and seek medical treatment in tertiary hospitals will be selected.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum and urine iodine levels | 1 year from enrollment
TNM staging of papillary thyroid cancer | 3 month from enrollment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi JY, Lee JH, Song Y. Evaluation of Iodine Status among Korean Patients with Papillary Thyroid Cancer Using Dietary and Urinary Iodine. Endocrinol Metab (Seoul). 2021 Jun;36(3):607-618. doi: 10.3803/EnM.2021.1005. Epub 2021 Jun 21. PMID 34154044
- [Background] Kim HJ, Park HK, Byun DW, Suh K, Yoo MH, Min YK, Kim SW, Chung JH. Iodine intake as a risk factor for BRAF mutations in papillary thyroid cancer patients from an iodine-replete area. Eur J Nutr. 2018 Mar;57(2):809-815. doi: 10.1007/s00394-016-1370-2. Epub 2017 Mar 3. PMID 28258306
- [Background] Zhang X, Zhang F, Li Q, Aihaiti R, Feng C, Chen D, Zhao X, Teng W. The relationship between urinary iodine concentration and papillary thyroid cancer: A systematic review and meta-analysis. Front Endocrinol (Lausanne). 2022 Oct 31;13:1049423. doi: 10.3389/fendo.2022.1049423. eCollection 2022. PMID 36387866
- [Background] Kim K, Cho SW, Park YJ, Lee KE, Lee DW, Park SK. Association between Iodine Intake, Thyroid Function, and Papillary Thyroid Cancer: A Case-Control Study. Endocrinol Metab (Seoul). 2021 Aug;36(4):790-799. doi: 10.3803/EnM.2021.1034. Epub 2021 Aug 11. PMID 34376043
- [Background] Lee JH, Hwang Y, Song RY, Yi JW, Yu HW, Kim SJ, Chai YJ, Choi JY, Lee KE, Park SK. Relationship between iodine levels and papillary thyroid carcinoma: A systematic review and meta-analysis. Head Neck. 2017 Aug;39(8):1711-1718. doi: 10.1002/hed.24797. Epub 2017 May 17. PMID 28513893